CLINICAL TRIAL: NCT05038943
Title: Evaluation of Safety and Effectiveness of The Paragonix™ SherpaPak Cardiac Transport System in Donation After Circulatory Death Heart Transplantation
Brief Title: Evaluation of Safety and Effectiveness of The SherpaPak in Donation After Circulatory Death Heart Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 0478-21-FB
Record Dates: First submitted 2021-08-31; First posted 2021-09-09 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Heart Transplant Failure; Determination of Death; Outcomes Research; Extracorporeal Membrane Oxygenation
Keywords: Transplantation, heart; Normothermic Regional Perfusion; Organ transport
MeSH Terms: conditions — Death

STUDY DESIGN:
Intervention Model Description: Cardiac allografts recovered from donors after circulatory death with thoracoabdominal normothermic regional perfusion will be transported with Paragonix SherpaPak Cardiac Transport System to the recipient center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SherpaPak (Experimental): cardiac allografts recovered from donors after circulatory determined death using thoracoabdominal normothermic regional perfusion will be transported to the recipient center in Paragonix SherpaPak Cardiac Transport System
  Interventions: Device: Paragonix SherpaPak Cardiac Transport System

INTERVENTIONS:
Device: Paragonix SherpaPak Cardiac Transport System — Transportation of cardiac allografts in a device maintaining constant optimal temperature to minimize freezing tissue injury

SUMMARY:
This is a prospective, pilot trial to evaluate the safety and effectiveness of The Paragonix SherpaPak™ Cardiac Transport System ("SherpaPak CTS") in transportation of cardiac allografts recovered from donors after circulatory death with thoracoabdominal normothermic regional perfusion (TA-NRP). SherpaPak™ CTS is an ultraportable hypothermic preservation and transport system that has been approved by United States Food & Drug Administration (FDA) for clinical use in heart transplantation.

DETAILED DESCRIPTION:
The investigators will accept donors between the ages of 18 and 49 without any known history of coronary artery disease, insulin dependent diabetes, or long-term smoking (>20 pack/years) and normal baseline cardiac function (EF>50) assessed with transthoracic echocardiogram. Donors will be selected and matched to the recipients based on standard criteria (blood group, cross-match, size match, and clinical stability). The current procedure of donation after circulatory death (DCD) and procurement follows a well-established course. After consent is obtained, the organs are allocated through United Network for Organ Sharing (UNOS). All organs will be recovered with protocolized UNMC DCD TA-NRP technique that involves reestablishment of blood flow in-situ after donor's circulatory arrest using portable venoarterial extracorporeal membrane oxygenation (VA-ECMO). Organs will be transported from a donor site to recipient center with the SherpaPak™ CTS. All organs will be transplanted at Nebraska Medicine. Recipients ("subjects") will be followed from transplant through one-year post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Recipient is ≥ 19 years old
2. Recipient, or their designated healthcare proxy, is able and willing to sign informed consent
3. Recipient meets standard listing criteria for heart transplantation

Exclusion Criteria:

1. Recipient is < 19 years old
2. Recipient, or their designated healthcare proxy, is unable to sign informed consent
3. Recipient has any condition that, in the opinion of the Investigator, would make study participation unsafe or would interfere with the objectives of the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Primary Graft Dysfunction (PGD) | 72 hours
  PGD will be classified according to International Society for Heart and Lung Transplantation (ISHLT) classification into: PGD-LV Grade 1 (LVEF ≤ 40% by echocardiography, or Hemodynamics with RAP > 15 mm Hg, PCWP > 20 mm Hg, CI < 2.0 L/min/m2 (lasting more than 1 hour) requiring low-dose inotropes); PGD-LV Grade 2 (I. One criteria from the following: Left ventricular ejection fraction ≤ 40%, or Hemodynamic compromise with RAP > 15 mm Hg, PCWP > 20 mm Hg, CI < 2.0 L/min/m2, hypotension with MAP < 70 mm Hg (lasting more than 1 hour) II. One criteria from the following: High-dose inotropes-Inotrope score >10, or Newly placed IABP (regardless of inotropes)); PGD-LV Grade 3 ( Dependence on left or biventricular mechanical support including ECMO, LVAD, BiVAD, or percutaneous LVAD. Excludes requirement for IABP; PGD-RV (I. Hemodynamics with RAP > 15 mm Hg, PCWP < 15 mm Hg, CI < 2.0 L/min/m2, II. TPG < 15 mm Hg and/or pulmonary artery systolic pressure < 50 mm Hg, III. Need for RVAD)

SECONDARY OUTCOMES:
Need for cardioversion or pacing to restart transplanted heart | 72 hours
  Need for cardioversion or pacing to restart transplanted heart
Vasoactive-inotropic score (VIS) | 24, 48, and 72 hours
  The vasoactive-inotropic score (VIS) will be calculated as a weighted sum of all administered inotropes and vasoconstrictors, reflecting pharmacological support of the cardio-vascular system. Formula for VIS calculation: dopamine dose (µg/kg/min) + dobutamine dose (µg/kg/min) + 100 x epinephrine dose (µg/kg/min) + 100 x norepinephrine dose (µg/kg/min).
Duration of vasoactive-inotropic support in days | 1 year
  Duration of vasoactive-inotropic support in days
Intensive Care Unit & Hospital length of stay in days | 1 year
  Intensive Care Unit & Hospital length of stay in days
Survival at discharge | 1 year
  Survival at discharge 30-day, 90-day, 1-year

CONTACTS AND LOCATIONS:
Overall Officials: Marian Urban, MD, PhD, Principal Investigator — Assistant Professor
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Radakovic D, Karimli S, Penov K, Schade I, Hamouda K, Bening C, Leyh RG, Aleksic I. First clinical experience with the novel cold storage SherpaPak system for donor heart transportation. J Thorac Dis. 2020 Dec;12(12):7227-7235. doi: 10.21037/jtd-20-1827. PMID 33447411
- [Result] Toldo S, Quader M, Salloum FN, Mezzaroma E, Abbate A. Targeting the Innate Immune Response to Improve Cardiac Graft Recovery after Heart Transplantation: Implications for the Donation after Cardiac Death. Int J Mol Sci. 2016 Jun 17;17(6):958. doi: 10.3390/ijms17060958. PMID 27322252
- [Result] Kobashigawa J, Zuckermann A, Macdonald P, Leprince P, Esmailian F, Luu M, Mancini D, Patel J, Razi R, Reichenspurner H, Russell S, Segovia J, Smedira N, Stehlik J, Wagner F; Consensus Conference participants. Report from a consensus conference on primary graft dysfunction after cardiac transplantation. J Heart Lung Transplant. 2014 Apr;33(4):327-40. doi: 10.1016/j.healun.2014.02.027. Epub 2014 Mar 5. PMID 24661451
- [Result] Yamazaki Y, Oba K, Matsui Y, Morimoto Y. Vasoactive-inotropic score as a predictor of morbidity and mortality in adults after cardiac surgery with cardiopulmonary bypass. J Anesth. 2018 Apr;32(2):167-173. doi: 10.1007/s00540-018-2447-2. Epub 2018 Jan 13. PMID 29332153